CLINICAL TRIAL: NCT02187185
Title: Studies of Salivary Inflammatory Biomarkers During Biofilm Overgrowth: Confirmation of Predictors and Comparative Effects of Sonicare/Elite-Flexcare in Various Stages of Periodontal Disease
Brief Title: Salivary Inflammatory Biomarkers: Predictors & Comparative Effects of Sonicare/Elite-Flexcare in Stages of Perio Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Philips Oral Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 09-0627
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2017-01

CONDITIONS: Inflammation; Periodontitis
Keywords: Inflammatory biomarkers; Periodontitis
MeSH Terms: conditions — Inflammation; Periodontitis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sonicare Elite-Flexcare (Active Comparator): Arm 1 participants will abstain from brushing and flossing teeth in selected sites which will typically be one maxillary and mandibular posterior sextant during a three week, no-hygiene phase via placement of acrylic stents. After the stent-induced biofilm overgrowth (SIBO) induction, the resolution phase of the study will involve a randomization that places half of the subjects on the Sonicare/Elite/Flexcare toothbrush. Thus, the resolution phase is a RCT designed to treat SIBO in subjects with varying levels of disease. Participants will reinstate normal full mouth oral hygiene and daily plaque control, exclusive of flossing, with dispensed dentifrice and toothbrush. Participants will be followed for four weeks during SIBO resolution.
  Interventions: Other: Sonicare/Elite-Flexcare Toothbrush
- Manual Toothbrush (Active Comparator): Arm 2 participants will abstain from brushing and flossing teeth in selected sites which will typically be one maxillary and mandibular posterior sextant during a three week, no-hygiene phase via placement of acrylic stents. After the stent-induced biofilm overgrowth (SIBO) induction, the resolution phase of the study will involve a randomization that places half of the subjects on the manual toothbrush. Thus, the resolution phase is a RCT designed to treat SIBO in subjects with varying levels of disease. Participants will reinstate normal full mouth oral hygiene and daily plaque control, exclusive of flossing, with dispensed dentifrice and toothbrush. Participants will be followed for four weeks during SIBO resolution.
  Interventions: Other: Manual Toothbrush

INTERVENTIONS:
Other: Sonicare/Elite-Flexcare Toothbrush — Philips Oral Healthcare product - battery powered menchanic toothbrush with nylon bristles
  Arms: Sonicare Elite-Flexcare
Other: Manual Toothbrush — traditional (non-mechanical) toothbrush with nylon bristles and plastic handle
  Arms: Manual Toothbrush

SUMMARY:
This research study has 2 aims. One aim is to see if saliva testing can show if a person has healthy gum tissue, gingivitis, or one of three degrees of periodontitis - mild, moderate, or severe. The second aim is to examine the effect of the Sonicare Elite/Flexcare toothbrush on periodontitis.

DETAILED DESCRIPTION:
Randomized controlled trial to determine clinical and inflammatory benefits of Sonicare Flexcare tooth brushing following experimental induction of biofilm overgrowth in various periodontal conditions.

This research study has both a Diagnostic Aim and a Treatment Aim. Aim #1 is to examine the utility of candidate inflammatory biomarkers within saliva to discriminate between health, gingivitis, mild, moderate and severe periodontis; and to discriminate between active versus inactive states of periodontal disease to see if these basal levels can predict the clinical response to biofilm overgrowth among various periodontal conditions; Aim #2 is to extend the claim of the anti-inflammatory and anti-infective efficacy of the Sonicare/Elite-Flexcare as compared to manual brushing to include 4 levels of periodontal disease [BGI-G, P1, P2 and P3].

The devices used in this study are subject only to Class I (general controls) and considered exempt from the premarket notification procedures and not subject to section 510(k), 515, or 520(m,) of the FDC Act in order to be legally marketed. Thus, the study does not meet the definition of an Applicable Clinical Trial.

ELIGIBILITY:
Inclusion Criteria:

1. adult males or females between the ages of 18 and 75 years (inclusive).
2. able and willing to follow study procedures and instructions.
3. read, understood and signed an informed consent form.
4. present with at least 8 teeth in the functional dentition with a minimum of 3 adjacent teeth with interproximal papilla in each posterior sextant that will have the stent.
5. be in good general health.
6. present with one of the following five categories to be considered for enrollment

   * BGI health (all PD<3mm, BOP<10%)
   * BGI-gingivitis (all PD≤3mm, BOP≥10%)
   * BGI-P1 (1+ site with PD>3mm, BOP≤10%)
   * BGI-P2 (1+ site with PD>3mm, BOP>10% but BOP≤50%)
   * BGI-P3 (1+ site with PD>3mm, BOP>50%)

Exclusion Criteria:

1. chronic disease with oral manifestations or active infectious diseases such as hepatitis, HIV or tuberculosis.
2. gross oral pathology.
3. treatment with antibiotics for any medical or dental condition within 1 month prior to the screening examination.
4. chronic treatment (i.e., two weeks or more) with any medication known to affect periodontal status (e.g., phenytoin, calcium antagonists, cyclosporin, anticoagulants, non-steroidal anti-inflammatory drugs, high dose aspirin such as >100mg per day) within one month of the screening examination.
5. ongoing medications initiated less than three months prior to enrollment (i.e., medications for chronic medical conditions must be initiated at least three months prior to enrollment).
6. clinically significant organ disease including impaired renal function, and/or any bleeding disorder.
7. severe unrestored caries, or any condition that is likely to require antibiotic treatment during the study, including the need for prophylactic antibiotic.
8. use any tobacco products or who have used tobacco products within the previous six months of the screening examination.
9. pregnant, or expect to become pregnant within the next three months and individuals nursing.
10. dental appliances that will interfere with stent construction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2009-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in (inflammatory biomarkers?) among a range of periodontal disease groups after using Sonicare Elite/Flexcare versus manual toothbrush for four weeks. | Four weeks

SECONDARY OUTCOMES:
Identification of salivary biomarkers that can distinguish between and among the 5 disease categories (health, gingivitis, and 3 levels of periodontal disease). | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven Offenbacher, DDS PhD MMSc, Principal Investigator — The University of North Carolina at Chapel Hill School of Dentistry
Locations (1):
- The University of North Carolina at Chapel Hill School of Dentistry, Chapel Hill, North Carolina, United States